CLINICAL TRIAL: NCT03744286
Title: Investigation Into an Innovative, Clinical Slip Inducing Device in the Chronic Incomplete Spinal Cord Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Director Max Näder Center, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STU00207310
Record Dates: First submitted 2018-09-25; First posted 2018-11-16 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: This is a 2-visit clinical trial to test a novel prototype slip inducing platform device for feasibility and not health outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Balance Slip (Experimental): * Perform standard clinical balance assessments
  * Determine the optimal slip distance by 10 passes each with plank movement of 2", 4", 6" and 8" on visit 1
  Interventions: Device: Slip Training

INTERVENTIONS:
Device: Slip Training — -On a separate day (visit 2), using the identified optimal distance, a training session that involves 24 passes on the device where 1-2 planks move will be performed.

SUMMARY:
The objective of this project is to fully test a newly developed affordable cost variable slip inducer in the ambulatory, incomplete spinal cord population. It is a self-contained device using a moving serial plank mechanism with wheels on the underside of each plank that allow for structured slips while a person walks over the planks with a harness for safety.

DETAILED DESCRIPTION:
All planks appear the same but can be adjusted on the underside allowing for it to be stable or can allow a slip in the forward and/or backward direction of up to 8 inches. This distance was determined from a review of slip bio-mechanics that noted that a slip is likely to occur when a slip distance exceeds 10 cm (3.9 inches) with the probability of recovery decreasing as the distance increases. The first goal of the project is to determine the optimal distance required for individuals with incomplete spinal cord injuries to have a 50% fall rate, as healthy individuals were found to have a fall rate of 50% at 11 inches. Investigators will then look at common clinical assessments and examine their ability to predict an individual's ability to recover from the individual's identified optimal slip distance. Investigators will also look at within session training effect on a person's balance control following a training session using the device.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a traumatic or non-traumatic incomplete spinal cord injury at least 6 months ago
* Between the ages of 18-85 years old.
* Ambulates as their primary means of mobility
* Able to walk without cane/crutch/walker for 30 feet.
* Weight less than 275 lbs.
* Medical clearance from physician

Exclusion Criteria:

* Uses a wheelchair as primary means of mobility
* Recent (<6 months) lower extremity fracture
* Other neurological diagnoses that would impact balance such as peripheral neuropathy, stroke, brain injury, etc.
* Lower extremity amputation
* Currently pregnant
* Uses knee-ankle-foot-orthosis for mobility.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Static Balance | Assessment Session 1 (baseline test, Will occur at the start of Visit 1, Day 1), Assessment Session 2 (conducted before Training during Visit 2, Day 2), Assessment Session 3 (Post Training Assessment; conducted at the end of Training Visit 2, Day 2)
  During the static stability test, the participants will be instructed to stand on the force plate as still as possible for 60 seconds with their eyes open. After 2 minutes of rest, the task will be repeated with the eyes closed. The excursions of the center of pressure (COP) and EMG of leg muscles will be analyzed.
  The AMTI Force System from Water Town, MA will be used to for this test. The platform is placed on the floor and subjects stand on the device. The force plate measures the forces and movements applied to its top surface.
Change in Dynamic Balance | Assessment Session 1 (baseline test, Will occur at the start of Visit 1, Day 1), Assessment Session 2 (conducted before Training during Visit 2, Day 2), Assessment Session 3 (Post Training Assessment; conducted at the end of Training Visit 2, Day 2)
  During the dynamic stability test, the ability to voluntarily displace the COP to a maximum distance without losing balance will be assessed (Limits of stability (LOS) test). The participant will be instructed to lean forward, backward, left, and right, hold the position for ~5 seconds and return back to the initial/center position.
  The AMTI Force System from Water Town, MA will be used to for this test.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No